CLINICAL TRIAL: NCT01302249
Title: A Phase 2, Double-masked, Randomized, Active-controlled, Crossover Study Assessing the Safety and Ocular Hypotensive Efficacy of AR-12286 or Timolol Added to Patients With Elevated Intraocular Pressure Currently Using Latanoprost
Brief Title: AR-12286 in Combination With Latanoprost
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aerie Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AR-12286-CS203
Record Dates: First submitted 2011-02-18; First posted 2011-02-24 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-04

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: Glaucoma; Intraocular pressure; Ocular hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AR-12286 (Experimental): AR-12286 Ophthalmic Solution 0.5%
  Interventions: Drug: Latanoprost 0.005%; Drug: AR-12286 Ophthalmic Solution 0.5%
- Timolol (Active Comparator): Timolol maleate ophthalmic solution 0.5%
  Interventions: Drug: Latanoprost 0.005%; Drug: Timolol maleate ophthalmic solution 0.5%

INTERVENTIONS:
Drug: Latanoprost 0.005% — q.d.
  Other Names: Xalatan(R)
Drug: AR-12286 Ophthalmic Solution 0.5%
  Arms: AR-12286
Drug: Timolol maleate ophthalmic solution 0.5%
  Arms: Timolol

SUMMARY:
This is a double-masked, randomized, multi-center, active-controlled, crossover comparison of the addition of AR-12286 or timolol to latanoprost in the treatment of elevated intraocular pressure (IOP).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or greater.
* Diagnosis of open angle glaucoma (OAG) or ocular hypertension (OHT).
* Currently using prostaglandin analogue (monotherapy or combination therapy) O.U. ≥ 1 month at time of study entry (first qualification visit) in study eye(s).
* Qualification Visit 1 (Screening) IOP at 16:00 hrs: PG monotherapy patients: ≥ 18 mm Hg; Combination therapy patients: >= 16 mm Hg. Qualification Visit 2 (post latanoprost run-in) IOP ≥ 20 mm Hg at 08:00 hrs and 10:00 hrs, IOP ≥ 18 mm Hg at 16:00 hrs in study eye(s). (Note: combination therapy may include any combination of topical ocular hypotensive agents).
* Corrected visual acuity in each eye +1.0 logMAR or better by ETDRS in each eye (equivalent to 20/200).
* Able and willing to give signed informed consent and follow study instructions

Exclusion Criteria:

In either eye:

* Previously randomized to treatment in a clinical study of AR-12286.
* Intraocular pressure > 36 mm Hg.
* History of acute angle-closure glaucoma, or closed or narrow angle upon gonioscopy
* Known hypersensitivity or contraindication to timolol maleate ophthalmic solution, or any component of the formulation (benzalkonium chloride, etc.), or to topical anesthetics, including history of conjunctival hyperemia with topical latanoprost of severity greater than 1 on a 0-3 scale.
* Ocular trauma within the past six months, or ocular surgery or laser treatment within the past three months.
* Contact lens wear within 30 minutes of instillation of study medication.
* PG monotherapy patients: Ocular hypotensive medication (other than prostaglandin) within 4 weeks of Visit 0 (Study entry, first qualification visit). Combination therapy patients: Ocular hypotensive medication (other than prostaglandin and current additional agent) within 4 weeks of Visit 0 (Study entry, first qualification visit).
* Conjunctival hyperemia of grade 2+ or greater at Visit 1.
* Any other ocular medication within 4 weeks of Visit 1 with the exception of lubricating drops for dry eye (which may be used throughout the study).
* Clinically significant ocular disease (e.g. corneal edema, uveitis, severe keratoconjunctivitis sicca) which might interfere with the study, including glaucomatous damage so severe that treatment with only latanoprost for two periods of up to 4 weeks is not judged safe (e.g., advanced glaucomatous optic nerve head or visual field loss).
* Any abnormality preventing reliable applanation tonometry of either eye.

In study eye(s):

* Glaucoma: pseudoexfoliation or pigment dispersion component, history of angle closure. Note: Previous laser peripheral iridotomy is acceptable.
* Previous glaucoma intraocular surgery or laser procedures.
* Refractive surgery (e.g., radial keratotomy, PRK, LASIK, etc.).
* Central corneal thickness greater than 600 µ.

Systemic:

* Known bronchial asthma (history or current), severe chronic obstructive pulmonary disease, sinus bradycardia, second or third degree atrioventricular block or overt cardiac failure.
* Clinically significant abnormalities in laboratory tests at screening, recognizing that subjects are not fasting at the time of drawing blood.
* Clinically significant systemic disease (e.g., uncontrolled diabetes, myasthenia gravis, hepatic, renal, cardiovascular or endocrine disorders) which might interfere with the study.
* Participation in any investigational study within the past 30 days.
* Changes of systemic medication that could have a substantial effect on IOP 4 weeks prior to screening, or anticipated during the study.
* Women of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2011-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure | 28 days
  The primary efficacy endpoint will be the mean IOP across subjects within treatment group at each study visit at each post-treatment timepoint.

SECONDARY OUTCOMES:
Ocular safety | 28 days
  Safety endpoints will be visual acuity, objective biomicroscopic and ophthalmoscopic examination, and subjective comfort as measured by adverse events in response to subject symptom queries.
Systemic safety | 28 days
  Heart rate, and blood pressure.

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - David Silverstone, M.D., New Haven, Connecticut
  - Coastal Research Associates, LLC, Roswell, Georgia
  - Heart of America Eye Care, P.A., Shawnee Mission, Kansas
  - Taustine Eye Center, Louisville, Kentucky
  - Alan L Robin, M.D., Baltimore, Maryland
  - Comprehensive Eye Care, St Louis, Missouri
  - Rochester Ophthalmology Group, Rochester, New York
  - Glaucoma Consultants of the Capital Region, Slingerlands, New York
  - Thomas K. Mundorf, M.D., Charlotte, North Carolina
  - Charlotte Eye Ear Nose and Throat, Charlotte, North Carolina
  - The Eye Institute, Tulsa, Oklahoma
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Cataract & Glaucoma Center, El Paso, Texas
  - Stacy R. Smith, M.D., Salt Lake City, Utah